CLINICAL TRIAL: NCT02619643
Title: Primed vs Unprimed Facilitatory and Depressive Paired Associative Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Device Feasibility
Other Study IDs: 1601M82561
Record Dates: First submitted 2015-11-25; First posted 2015-12-02 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Healthy
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Primed PAS 1A (Experimental): Two sessions of paired associative stimulation (PAS) using transcranial magnetic stimulation will be applied consecutively (within minutes).
  Interventions: Device: Transcranial Magnetic Stimulation (Magstim)
- Unprimed PAS 1B (Experimental): A single session of active paired associative stimulation (PAS) using transcranial magnetic stimulation will be applied.
  Interventions: Device: Transcranial Magnetic Stimulation (Magstim)
- Sham PAS (Sham Comparator): A single session of sham paired associative stimulation (PAS) using transcranial magnetic stimulation will be applied
  Interventions: Device: Transcranial Magnetic Stimulation (Magstim)
- Primed PAS 2A (Experimental): Two sessions of paired associative stimulation (PAS) using transcranial magnetic stimulation will be applied consecutively (within minutes).
  Interventions: Device: Transcranial Magnetic Stimulation (Magstim)
- Unprimed PAS 2B (Experimental): A single session of active paired associative stimulation (PAS) using transcranial magnetic stimulation will be applied.
  Interventions: Device: Transcranial Magnetic Stimulation (Magstim)
- Primed PAS 1C (Experimental): Two sessions of paired associative stimulation (PAS) using transcranial magnetic stimulation will be applied consecutively (within minutes).
  Interventions: Device: Transcranial Magnetic Stimulation (Magstim)
- Primed PAS 2C (Experimental): Two sessions of paired associative stimulation (PAS) using transcranial magnetic stimulation will be applied consecutively (within minutes).
  Interventions: Device: Transcranial Magnetic Stimulation (Magstim)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (Magstim)
  Other Names: TMS; Magstim

SUMMARY:
Following brain injury (e.g. stroke), application of non-invasive brain stimulation may improve rehabilitative efforts. However, the most effective method of non-invasive brain stimulation is unknown. Paired associative stimulation (PAS) is a method of non-invasive brain stimulation that pairs an electrical peripheral nerve stimulus with a magnetic stimulus to the head. This method can be applied in a manner that increases (facilitates) or decreases (depresses) excitability within the brain. Furthermore, applying two consecutive PAS sessions within minutes of each other (called primed PAS) may augment changes in excitability more than a single PAS session alone.

Thus, the purpose of this study is to compare the effect of a double PAS session (primed PAS) to the effect of a single PAS session (unprimed PAS) and a sham PAS session in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 30 years of age
* Elicitable motor evoked potential from the motor cortex contralateral to the dominant hand
* Elicitable N20 sensory evoked potential

Exclusion Criteria:

* History of neurological disease
* Seizure within the past 2 years
* Currently taking epileptogenic medication
* Peripheral neuropathy
* Cognitive impairment and/or major psychiatric disorder
* Metal in the head (dental permitted)
* Pacemaker or other indwelling devices
* Pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline peak-to-peak amplitude of motor evoked potential | Immediately before and within 60 minutes following intervention
  Single-pulse TMS will be used to evoke a motor response that is recorded using electromyography (EMG). The peak-to-peak amplitude of the EMG response will be measured.
Change from baseline resting motor threshold | Immediately before and within 60 minutes following intervention
  Single-pulse TMS will be used to evoke a motor response that is recorded using electromyography (EMG). The lowest stimulator output needed to elicit a consistent response will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Frost, MS, Principal Investigator — University of Minnesota